CLINICAL TRIAL: NCT05710367
Title: Effects Of Sodium Glucose Cotranspoter 2 Inhibitors On Heart And Kidneys In Fabry Disease Patients; A Prospective, Randomized, Double-Blind, Placebo- Controlled Study.
Brief Title: Effects Of Sodium Glucose Cotranspoter 2 Inhibitors On Heart And Kidneys In Fabry Disease Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Albina Nowak, MD (Other)
Responsible Party: Sponsor-Investigator, Albina Nowak, MD, Principal Investigator, Senior Physician of Endocrinology, Diabetes and Clinical Nutrition, University of Zurich
Organization: University of Zurich (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SGLT2Is46
Record Dates: First submitted 2023-01-10; First posted 2023-02-02 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-01

CONDITIONS: Fabry Disease
MeSH Terms: conditions — Fabry Disease | interventions — dapagliflozin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dapagliflozin 10mg Tab (Experimental): SGLT2is- Dapagliflozin (Forxiga): 10 mg/d, oral drug
  Interventions: Drug: Dapagliflozin 10mg Tab
- Placebo (Placebo Comparator): Placebo tablet will have the same color, taste, smell and package as the verum tablet
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dapagliflozin 10mg Tab — Forxiga® as an add-on treatment in patients with renal and/or cardiac association FD in an exploratory framework.
  Arms: Dapagliflozin 10mg Tab
Drug: Placebo — matched oral drug. Placebo tablet will have the same color, taste, smell and package as the verum tablet
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to test dapagliflizone in Fabry patients. The main questions it aims to answer are:

* Has 10 mg/d of dapagliflozin a positive effect on kidney functions of Fabry patients.
* Has 10 mg/d of dapagliflozin a positive effect on heart functions in Fabry patients.

Participants will be asked to

* Sign an informed consent
* Give a blood and urine samples
* Be subjected to Echocardiography investigation
* Take 10 mg/day Dapagliflizone

Researchers will compare treatment to placebo groups to see if kidneys and heart functions will be improved in the treatment group better more than the placebo group.

ELIGIBILITY:
Inclusion Criteria

* Age: 18-70 years
* Patients with genetically confirmed Fabry disease.
* On treatment with Enzyme Replacement Therapy (ERT).
* ERT or chaperone therapy at stable dose for at least 3 last months
* Albuminuria >35 mg/day and/or proteinuria >150 mg/day
* eGFR ≥25 mL/min/1.73 m2
* On a stable dose of an ACEi, ARB or renin receptors blockers for at least 4 weeks prior to randomization
* Sufficient command of German language.
* Signed and dated informed consent.
* Known cardiac association of FD

Exclusion Criteria:

* Known hypersensitivity, allergy or contraindications to dapagliflozin.
* Diagnosis of type 1 or type 2 diabetes mellitus
* Patients with any disease (other than Fabry disease) affecting the heart and the kidnys.
* History of kidney transplantation.
* Active malignancy.
* Use of the co-interventional treatments (Aldosterone antagonists, Continuous use of NSAIDs or systemic steroids) within 6 weeks of screening will not be allowed.
* Any medication, surgical or medical condition which might significantly alter the absorption, distribution, metabolism, or excretion of medications including, but not limited to any of the following:

  1. History of active inflammatory bowel disease within the last six months;
  2. Major gastrointestinal tract surgery such as gastrectomy, gastroenterostomy, or bowel resection;
  3. Gastro-intestinal ulcers and/or gastrointestinal or rectal bleeding within last six months;
  4. Pancreatic injury or pancreatitis within the last six months;
  5. Evidence of hepatic disease as determined by any one of the following: ALT or AST values exceeding 3x ULN at the screening visit, a history of hepatic encephalopathy, a history of esophageal varices, or a history of portocaval shunt;
* Subject who, in the assessment of the investigator, may be at risk for dehydration or volume depletion that may affect the interpretation of efficacy or safety data.
* Donation or loss of 400 mL or more of blood within 8 weeks prior to initial dosing.
* Any surgical or medical condition, which in the opinion of the investigator, may place the patient at higher risk from his/her participation in the study, or is likely to prevent the patient from complying with the requirements of the study or completing the study.
* Women who are pregnant or breast feeding; intention to become pregnant during the course of the study, lack of safe contraception.
* Patients with known or suspected non-compliance, drug or alcohol abuse, including Marijuana cigarettes.
* Participation in another study with investigational drugs within the 30 days preceding and during the present study.
* Enrolment of the investigator, his/her family members, employees and other dependent persons.
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Assess the change of eGFR in treatment months 6, 12 and at baseline | Baseline, 6 months and 12 months
  The CKD-EPI (Chronic Kidney Disease Epidemiology Collaboration) 2009 formula are used to evaluate the calculated GFR.
  eGFR in month 6 and 12 are compared to baseline eGFR.
Assess the change of Protein /creatinine ratio in urine | Baseline, 6 months and 12 months
  Total protein is measured in the morning sample of urine, minimal volume of 10 ml are collected and analyzed using Immune nephelometry method. Protein concentration are reported in relation to creatinine.
Assess the change of Albumin/creatinine ratio in urine | Baseline, 6 months and 12 months
  Albumin is measured in the morning sample of urine, minimal volume of 10 ml are collected and analyzed using Immune nephelometry method. Albumin concentration are reported in relation to creatinine.

SECONDARY OUTCOMES:
NT-pro BNP level will be assessed at baseline and after 6 and 12 months of treatment with study drug and placebo | Baseline, 6 months and 12 months
  NT-pro BNP are assessed using a minimal of 2.5 ml heparin-plasma sample with Electro- Chemiluminescent Immunoassay technique.
Troponin I levels will be assessed at baseline and after 6 and 12 months of treatment with | Baseline, 6 months and 12 months
  Troponin I are measured in heparin whole blood (min. 2.5 ml) using Chemiluminescent Microparticle Immunoassay.
LVMMI parameter will be assessed at baseline and after 6 and 12 months of treatment with study drug and placebo | Baseline, 6 months and 12 months
  LVMMI parameter are assessed using M-mode echocardiography in Cardiology clinic
Septal thickness parameter will be assessed at baseline and after 6 and 12 months of treatment with study drug and placebo | Baseline, 6 months and 12 months
  Septal thickness parameter are assessed using M-mode echocardiography in Cardiology clinic

OTHER OUTCOMES:
Chlosterol level will be assessed at baseline and after 6 and 12 months of treatment with study drug and placebo | Baseline, 6 months and 12 months
  Chlosterol level are measured using a minimal of 2.5 ml heparin-plasma sample with Enzymatic color test (CHOD-POD method)

IPD SHARING:
Plan to Share IPD: Undecided